CLINICAL TRIAL: NCT02950376
Title: Development of Virtual Reality-Based Addiction Assessment System for Synthetic Drugs Addiction
Brief Title: The Novel Addiction Assessment Study in Synthetic Drugs Addiction
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Min ZHAO, Vice President, Shanghai Mental Health Center
Other Study IDs: MZhao-006
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Amphetamine Addiction
Keywords: synthetic drugs; virtual reality; addiction evaluation; physiological data; eye movement index
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group1：amphetamine abusers
  Interventions: Other: DSM-5 +Virtual reality-based addiction assessment system
- Group2: health control
  Interventions: Other: Virtual reality-based addiction assessment system
- Group3: norm of assessment system
  Interventions: Other: DSM-5 +Virtual reality-based addiction assessment system

INTERVENTIONS:
Other: DSM-5 +Virtual reality-based addiction assessment system — The patients who used the amphetamine type stimulants will be diagnosed by the chief physician、associate chief physician or attending physician first to evaluate their addiction severity. And then the patients will finish the test in the virtual environment, at the same time their eye movement index and other physiological data will be recorded .Physiological data includes cardiac rate、galvanic skin response and electroencephalogram and so on.The test will proceed at the beginning of withdrawl、3 months later、 6 months later and 1 year later and record the information synchronously.
  Groups: Group1：amphetamine abusers
Other: Virtual reality-based addiction assessment system — The healthy controls will finish the test in the virtual environment, at the same time their eye movement index and other physiological data will be recorded .Physiological data includes cardiac rate、galvanic skin response and electroencephalogram and so on.The test will proceed at the baseline and 1 month later and record the information synchronously.
  Groups: Group2: health control
Other: DSM-5 +Virtual reality-based addiction assessment system — The patients who used the amphetamine type stimulants will be diagnosed by the chief physician、associate chief physician or attending physician first to evaluate their addiction severity. And then the patients will finish the test in the virtual environment, at the same time their eye movement index and other physiological data will be recorded .Physiological data includes cardiac rate、galvanic skin response and electroencephalogram and so on.In this group which is designed to construct the norm of assessment system, the test will record the information synchronously and proceed after baseline assessment.
  Groups: Group3: norm of assessment system

SUMMARY:
The purpose of this research is to develop an objective assessment based on the virtual reality techniques which is used for evaluate addiction severity.

DETAILED DESCRIPTION:
In order to evaluate the addiction severity and the effect of rehabilitation objectively, this study develops a virtual environment model based on the virtual reality technique, making the subjects in a drug related or neutral scene , at the same time recording the physical signs and eye movements index. Reliability and validity of this system will also be tested in this study. And we will construct the norm of addiction assessment system in Shanghai .The evaluating system will be very beneficial to develop novel and practical assessment for synthetic durg related disorder, and provide a reference for other drug dependence diagnosis.

ELIGIBILITY:
Criteria for synthetic drug abusers:

Inclusion Criteria:

* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-4) for methamphetamine (MA) use disorders;
* Education level equal or more than 9 years;
* Have normal or corrected-to-normal vision;
* Have normal or corrected-to-normal hearing;
* Less than 3 months before last drug use;

Exclusion Criteria:

* Current substance use (except nicotine or caffeine) ;
* History of disease which influence cognition，such as seizure disorder、cerebrovascular disease、 head injury or other severe medication conditions;
* Intelligence quotient less than 70.

Criteria for healthy control:

Inclusion Criteria:

* Without schizophrenia family history;
* Without history of drug abuse;
* Education level equal or more than 9 years;
* Have normal or corrected-to-normal vision;
* Have normal or corrected-to-normal hearing.

Exclusion Criteria:

* History of disease which influence cognition，such as seizure disorder、cerebrovascular disease、head injury or other severe medication conditions;
* Intelligence quotient less than 70.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study includes the synthetic drug abusers and healthy control into the experiment.The drug abusers will be recruited from compulsory isolated detoxification centers and non compulsory isolated detoxification institutions.The healthy control will be recruited from the residential communities.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes of physiological indexs | In 1 year
  The physiological index including galvanic skin response、encephlogram and electromyogram will be used to evaluate the reliability and validity of the virtual reality based addiction assessment system, and construct the norms of assessment system as well.
Changes of eye movement index | In 1 year
  The eye movement index will be used to evaluate the reliability and validity of the virtual reality based addiction assessment system, and construct the norms of assessment system as well.

SECONDARY OUTCOMES:
The Diagnostic and Statistical Manual of Mental Disorders（DSM） | baseline
  To establish the criterion validity
Addiction Severity Index(ASI) | baseline
  To establish the criterion validity

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No